CLINICAL TRIAL: NCT03821662
Title: Occupational Therapy Led Interdisciplinary Diabetes Self-Management Program
Brief Title: OT-Led Interdisciplinary Diabetes Self-Management Prgm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Hand Therapy Partners (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00009334
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus
Keywords: Diabetes; Occupational Therapy; Interdisciplinary Teams; Diabetes Self-Management Education (DSME); Diabetes Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OT Diabetes Self-Management Intervention (Experimental): The intervention is organized into five modules. Each participant receives an individually tailored combination of modules, and treatment activities within each module, as established through collaborative goal setting between the participant and OT during the initial evaluation. The five modules are: (1) Living with Diabetes-addressing gaps in the knowledge and skills necessary to effectively manage diabetes; (2) Access and Advocacy-strategies to collaborate and communicate with healthcare providers; (3) Activity and Health-analyzing daily habits and routines; (4) Social Support-strategies to address diabetes care in various social environments and to identify sources of support; (5) Emotional Well-Being-strategies to address stress, diabetes burnout, and depression.
  Interventions: Behavioral: OT Diabetes Self-Management Intervention

INTERVENTIONS:
Behavioral: OT Diabetes Self-Management Intervention — Occupational therapy chronic disease self-management intervention.

SUMMARY:
This study proposes to introduce an outpatient Occupational Therapy (OT)-led diabetes intervention program. OTs with training in diabetes self-management modules that address physical, social, emotional, and systemic factors that influence health. Patients receiving outpatient OT services for development of diabetes self-management skills will be seen for approximately 8 forty five-minute to one-hour sessions over 6 months. OTs will communicate with other interdisciplinary care team members using Electronic Health Record (EHR) messaging, phone calls, and in-person communication as needed. There will be at minimum a monthly consult meeting with a doctor of psychology (Psy D), registered dietitian (RD), social worker (SW), and pharmacist (PharmD), and the primary care medical team will be provided with monthly progress notes. The investigators hypothesize that participants demonstrate improved blood sugar levels, improved ability to take medications as directed, increases in overall sense of physical, mental, and social health, and positive changes in their self-efficacy related to diabetes self-management. The investigators also hypothesize that OT visits will be reimbursed by insurers more than 50% of all billed visits.

DETAILED DESCRIPTION:
Effective interventions to support patients' diabetes management are urgently needed to curtail the growing financial and human cost of diabetes. However, sustainable solutions to this health challenge have been elusive due to the intrinsic and extrinsic barriers patients face when attempting to incorporate necessary health behaviors into their daily routines (e.g., dietary changes, physical activity, medication management, blood glucose monitoring, and stress management). The focus of occupational therapy (OT) is to work with patients within the context of their daily lives. OTs identify current patient roles (work, family, community), habits, and routines, then work with the patient to identify and address barriers to diabetes self-management within these aspects of their daily lives. Within OT, an intervention approach informed by Lifestyle Redesign (LR) has been shown to be effective at improving diabetes-related health outcomes among people with diabetes. This study proposes to introduce an OT- led diabetes intervention program into an outpatient OT clinic. The intervention is an interdisciplinary team approach as the intervention is informed and monitored by the interdisciplinary team members, who are part of the planning process, and who will participate in regular review of the intervention and the patient needs. With OT leading the team to address barriers to lifestyle modification, the primary care medical team will continue to oversee the overall health care of the patient. The OT will communicate regularly with the primary care team.

OTs with training in diabetes education will deliver the intervention to patients in the study within the course of their typical work day at the OT clinic. Treatment activities and materials will be delivered in English or Spanish, per patient preference as one of the OT interventionists is fluent in Spanish. Patients receiving OT services for development of diabetes self-management skills will be seen for approximately 8 forty five-minute to one-hour sessions over 6 months. OT notes will be maintained within the Electronic Health Record (EHR) as is standard practice at this clinic; the therapist will communicate with other interdisciplinary care team members using EHR messaging, phone calls, and in-person communication as needed. There will be at minimum a monthly consult meeting with a doctor of psychology (Psy D), registered dietitian (RD), social worker (SW), and pharmacist (PharmD), and the primary care medical team will be provided with monthly progress notes.

The intervention will be offered in a one-on-one direct therapy format. The intervention will focus on lifestyle modification strategies that will improve the patient's diabetes self-management skills. The intervention is organized into five modules that address:

* living with diabetes,
* strategies to communicate with healthcare providers to ensure patient needs are met,
* analyzing and modifying patient habits and routines to determine what changes they must make to manage their diabetes,
* identify and use social supports to help manage diabetes
* strategies to reduce stress and depression, improve emotional well-being, and minimize risk of diabetes burn-out (patient frustration with living with the disease)

Each patient receives an individually tailored combination of modules, and treatment activities within each module as established through collaborative goal setting between the patient and OT during the initial evaluation.

The investigators will analyze outcomes using descriptive analytics and paired t-tests to test our hypotheses. The investigators will collect EHR data on HbA1c and compare pre/post measures of the clinically relevant self-report surveys on diabetes self care, and barriers to self-care and management (Diabetes Empowerment Scale, Medication Adherence Assessment Scale, and the Canadian Occupational Performance Measure), physical, mental, and social health (Patient-Reported Outcomes Measurement Information System® PROMIS-29). Changes in HbA1c levels will be tracked by obtaining recent levels from the patient's primary care team. With patients referred to the OT intervention who have not had an HbA1c within ≤4 weeks of the initial referral date, the OT will consult with the primary care physician and determine if an HbA1c level can be obtained as a part of their normal care. The investigators will collect EHR data on follow-up HbA1c testing scores that are available within 12 weeks of the 8th OT visit and self-report surveys the day of 8th OT visit. If a patient has completed the full intervention, the study staff will follow-up biweekly for no more than 3 months after their initial visit, and attempt to collect self-report data up to 6 months after the final visit to determine the sustainability of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Diabetes Mellitus Type 2
* Most recent HbA1c level >7.0% OR has been identified by medical provider as having uncontrolled diabetes
* English or Spanish Speaking
* Patient enrolled in a contracted commercial insurance plan or self-paying patients
* Expresses willingness to make lifestyle changes related to diabetes self-care

Exclusion Criteria:

* Patients that receive care through Workers Comp, or Motor Vehicle Insurance
* Patients that do not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Glycated hemoglobin (HbA1C) | Baseline & 6 months.
  Measure of blood glucose concentration over approximately the previous 12 weeks.

SECONDARY OUTCOMES:
Canadian Occupational Therapy Measure (COPM) | Baseline & 6 months.
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time. Areas of everyday living explored during the interview include self-care, productivity or leisure. The client is asked to rate the importance of each of the occupations to his/her life using a 10-point rating scale. Once the top five most important occupations are identified, the client is asked to use a 10 point scale to rate their own level of performance and satisfaction with performance for each of the five identified problems. The therapist calculates an average COPM performance score and satisfaction score. These typically range between 1 and 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction.
Change from Baseline Patient-Reported Outcomes Measurement Information SystemⓇ (PROMIS) 29 | Baseline & 6 months.
  29-item quality of life survey of self-reported physical, mental and social health and wellbeing. The seven 4-item subscales are comprised of 5-point Likert Scale questions. The subscales can be administered together or individually. There is also one 11-point rating scale for pain intensity. The total raw score is the sum the values of the response to each question. For the 4-item subscales the range of raw scores is 4-20. T-scores can be calculated by the PROMIScore computer program with our without missing responses.
Change from Baseline Diabetes Empowerment Scale (DES-SF) | Baseline & 6 months.
  8-item measure of the psychosocial self-efficacy of people with diabetes. An item checked "strongly agree" receives 5 points; "agree" - 4 points; "neutral" - 3 points; "disagree" - 2 points; and "strongly disagree" receives 1 point. The numerical values for a set of items in a particular subscale (for example: items 5-14 in the "Goal Setting" subscale) are added and the total is divided by the number of items (in this case 10) in the subscale. The resulting value is the score for that subscale. An overall score for the DES can be calculated by adding all of the item scores and dividing by 28.
Change from Baseline Medication Adherence Assessment Scale | Baseline & 6 months.
  A 7-item survey of self-reported medication adherence. Total raw score is the sum of all likert scale items ranging from 0-28 total points. Lower scores indicate better adherence than higher scores. A score of zero indicates good adherence for self-management. Scores greater than 2 for any item indicate the need for intervention to address barriers to medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Dahl-Popolizio, DBH, OTR/L, Principal Investigator — Arizona State University
Locations (1):
- Hand Therapy Partners, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark., F A, Blanchard., J, Sleight, A., Cogan, A., Florindez, L., Gleason, S.,…Vigen, C. (2015). Lifestyle redesign: The intervention tested in the USC well elderly studies (2nd ed.). AOTA Press: MD
- [Background] Pyatak EA, Carandang K, Vigen CLP, Blanchard J, Diaz J, Concha-Chavez A, Sequeira PA, Wood JR, Whittemore R, Spruijt-Metz D, Peters AL. Occupational Therapy Intervention Improves Glycemic Control and Quality of Life Among Young Adults With Diabetes: the Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) Randomized Controlled Trial. Diabetes Care. 2018 Apr;41(4):696-704. doi: 10.2337/dc17-1634. Epub 2018 Jan 19. PMID 29351961